CLINICAL TRIAL: NCT05448859
Title: The Effect of Oocyte Denudation Time and Intracytoplasmic Sperm Injection Time on Embryo Quality at Assisted Reproductive Technology Clinic
Brief Title: Effect of Oocyte Denudation Time and Intracytoplasmic Sperm Injection Time on Embryo Quality
Status: Completed | Type: Observational
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Other Study IDs: OBGY-202206.02
Record Dates: First submitted 2022-06-20; First posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Fertility Disorders
Keywords: infertility; assisted reproductive technology; embryo quality; oocyte denudation; intracytoplasmic sperm injection
MeSH Terms: conditions — Infertility | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 3-4 hours denudation: oocytes with 3-4 hours denudation time
  Interventions: Procedure: intracytoplasmic sperm injection
- 4-5 hours denudation: oocytes with 4-5 hours denudation time
  Interventions: Procedure: intracytoplasmic sperm injection
- 5-6 hours denudation time: oocytes with 5-6 hours denudation time
  Interventions: Procedure: intracytoplasmic sperm injection
- 6-7 hours denudation time: oocytes with 6-7 hours denudation time
  Interventions: Procedure: intracytoplasmic sperm injection
- more than 7 hours denudation time: oocytes with more than 7 hours denudation time
  Interventions: Procedure: intracytoplasmic sperm injection

INTERVENTIONS:
Procedure: intracytoplasmic sperm injection — injection of sperm into an oocyte in assisted reproductive technology
  Other Names: ICSI

SUMMARY:
An observational analytic retrospective study was conduct using cross-sectional study. The subject were oocytes from in-vitro fertilization procedures using the ICSI method at the assisted reproductive technology clinic in a private hospital in Bandung for the period 2017 - 2019. Three variables were oocyte denudation time, ICSI time and embryo quality collected from samples that met the research criteria.

DETAILED DESCRIPTION:
This study analyses the different oocyte denudation time after ICSI on all embryos generated during IVF procedures between 1 Januaryr 2017 and 31 December 2019. All oocytes arer categorised on how many hours their denudation times were and these were then assessed for their qualities.

ELIGIBILITY:
Inclusion Criteria:

* oocytes collected from in-vitro fertilisation procedures involving intracytoplasmic sperm injection

Exclusion Criteria:

* oocytes from patients >40 years old
* oocytes from primary infertility >5 years
* endometriosis
* polycystic ovarian syndrome

Ages: 3 Hours to 8 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Oocytes are derived from patients enrolled in IVF
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Oocyte denudation time | 3 hours
  time measured for oocyte denudation

CONTACTS AND LOCATIONS:
Overall Officials: Dian Tjahyadi, Principal Investigator — Universitas Padjadjaran

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised data on oocytes and IVF procedures are only available upon reasonable written request to the authors team.

REFERENCES:
- [Result] Isiklar A, Mercan R, Balaban B, Alatas C, Aksoy S, Urman B. Impact of oocyte pre-incubation time on fertilization, embryo quality and pregnancy rate after intracytoplasmic sperm injection. Reprod Biomed Online. 2004 Jun;8(6):682-6. doi: 10.1016/s1472-6483(10)61649-5. PMID 15169586